CLINICAL TRIAL: NCT03566940
Title: A Phase 2, Observer-blind, Active-controlled, Randomized Dose-finding Study in Healthy Infants to Assess the Safety, Reactogenicity and Immunogenicity of 3 Dose Levels of a Trivalent Inactivated Poliovirus Vaccine Based on Sabin Strains Compared to Conventional Salk IPV, in a 6, 10 and 14 Weeks of Age Immunization Schedule, and Co-administered With Diphtheria, Tetanus, Whole Cell Pertussis, Haemophilus Influenzae Type b, Hepatitis B, Pneumococcal Conjugate and Rotavirus Vaccines
Brief Title: A Study to Assess the Safety, Reactogenicity and Immunogenicity of a Trivalent Inactivated Poliovirus Vaccine (IPV) Based on Sabin Strains Compared to Conventional Salk IPV in a 6, 10 and 14 Weeks of Age Immunization Schedule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CR108472; GV000051POL2001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Low Dose IPV Based on Sabin Strains (sIPV) (Experimental): Participants will receive intramuscular (IM) injection of the low dose trivalent inactivated poliovirus vaccine (sIPV - 3 doses) at 6, 10 and 14 weeks of age. Participants will also be given a single booster vaccine of conventional Salk IPV (cIPV) at approximately 24 weeks after the third vaccination (38 weeks of age).
  Interventions: Biological: sIPV; Biological: cIPV
- Group 2: Intermediate Dose sIPV (Experimental): Participants will receive IM injection of the intermediate dose trivalent inactivated poliovirus vaccine (sIPV - 3 doses) at 6, 10 and 14 weeks of age. Participants will also be given a single booster vaccine of cIPV at approximately 24 weeks after the third vaccination (38 weeks of age).
  Interventions: Biological: sIPV; Biological: cIPV
- Group 3: High Dose sIPV (Experimental): Participants will receive IM injection of the high dose trivalent inactivated poliovirus vaccine (sIPV - 3 doses) at 6, 10 and 14 weeks of age. Participants will also be given a single booster vaccine of cIPV at approximately 24 weeks after the third vaccination (38 weeks of age).
  Interventions: Biological: sIPV; Biological: cIPV
- Group 4: Conventional Salk IPV (cIPV) (Active Comparator): Participants will receive IM injection of cIPV (3 doses) at 6, 10 and 14 weeks of age. Participants will also be given a single booster vaccine of cIPV at approximately 24 weeks after the third vaccination (38 weeks of age).
  Interventions: Biological: cIPV

INTERVENTIONS:
Biological: sIPV — Participants will receive 0.5 milliliter (mL) of sIPV as a solution for IM injection.
  Other Names: JNJ-64152348
  Arms: Group 1: Low Dose IPV Based on Sabin Strains (sIPV); Group 2: Intermediate Dose sIPV; Group 3: High Dose sIPV
Biological: cIPV — Participants will receive 0.5 mL of cIPV as a suspension for IM injection.

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of 3 different dose levels of inactivated poliovirus vaccine based on Sabin strains (sIPV) in healthy participants, using conventional Salk IPV (cIPV) as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Study participant is a boy or a girl, who is eligible for expanded programme on immunization (EPI) vaccinations (that is, inactivated poliovirus vaccine [IPV], Diphtheria, Tetanus, whole cell Pertussis [DTwP]-Haemophilus influenzae type b [Hib]-Hepatitis B virus [HBV] and 13-valent Pneumococcal conjugate vaccine [PCV13]) at Weeks 6, 10 and 14 and Rotavirus vaccination at Weeks 6 and 14
* Study participant has born after a normal term pregnancy (greater than or equal to [>=]37 weeks) and with a birth weight of >=2.5 kilogram (kg)
* Study participant must be healthy as confirmed by the investigator on the basis of physical examination, vital signs and medical history, including the course of the pregnancy and relevant medical history of the mother, such as but not limited to human immunodeficiency virus, Hepatitis B virus (HBV), hepatitis C virus status or other significant disease that might impact the participant's health. Information about the course of the pregnancy and relevant medical history of the mother is obtained from the mother in person and at the discretion of the investigator without the need for official documentation or testing
* Each study participant and his or her legally acceptable representative must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Study participant and his or her legally acceptable representative are available and reachable for all scheduled study visits and telephone contacts within the allowed window

Exclusion Criteria:

* Contraindication to intramuscular (IM) injections and blood draws (venipuncture) for example, bleeding disorders
* Known allergies, hypersensitivity, or intolerance to 1 of the excipients of IPV based on Sabin strains (sIPV) or conventional Salk IPV (cIPV) or any other vaccine component in the participant or mother
* Received polio vaccine or were previously infected with poliovirus
* Known or suspected autoimmune disease or persistent impairment/alteration of the immune function
* Known neurological disease including seizures, congenital defects, or genetic disorders (for example, Down syndrome)

Ages: 39 Days to 59 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Events (AEs) | 7 days after first vaccination
  Number of participants with solicited local and systemic AEs will be determined up to 7 days after first vaccination. Solicited local AEs (including erythema, swelling/induration, and pain/tenderness at the study vaccine injection site) and systemic AEs (loss of appetite/change in eating habits, vomiting, diarrhea, decreased activity/lethargy, increased or decreased sleep, irritability, persistent crying and fever) will be assessed.
Number of Participants with Solicited Local and Systemic AEs | 7 days after second vaccination
  Number of participants with solicited local and systemic AEs will be determined up to 7 days after second vaccination. Solicited local AEs (including erythema, swelling/induration, and pain/tenderness at the study vaccine injection site) and systemic AEs (loss of appetite/change in eating habits, vomiting, diarrhea, decreased activity/lethargy, increased or decreased sleep, irritability, persistent crying and fever) will be assessed.
Number of Participants with Solicited Local and Systemic AEs | 7 days after third vaccination
  Number of participants with solicited local and systemic AEs will be determined up to 7 days after third vaccination. Solicited local AEs (including erythema, swelling/induration, and pain/tenderness at the study vaccine injection site) and systemic AEs (loss of appetite/change in eating habits, vomiting, diarrhea, decreased activity/lethargy, increased or decreased sleep, irritability, persistent crying and fever) will be assessed.
Number of Participants with Unsolicited AEs | 28 days after first vaccination
  Number of participants with unsolicited AEs will be determined up to 28 days after first vaccination. Unsolicited AEs will include all AEs for which the participant's legally acceptable representative(s) is not specifically questioned in the participant diary. Unsolicited AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3), potentially life threatening (Grade 4), and death (Grade 5).
Number of Participants with Unsolicited AEs | 28 days after second vaccination
  Number of participants with unsolicited AEs will be determined up to 28 days after second vaccination. Unsolicited AEs will include all AEs for which the participant's legally acceptable representative(s) is not specifically questioned in the participant diary. Unsolicited AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3), potentially life threatening (Grade 4), and death (Grade 5).
Number of Participants with Unsolicited AEs | 28 days after third vaccination
  Number of participants with unsolicited AEs will be determined up to 28 days after third vaccination. Unsolicited AEs will include all AEs for which the participant's legally acceptable representative(s) is not specifically questioned in the participant diary. Unsolicited AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3), potentially life threatening (Grade 4), and death (Grade 5).
Number of Participants with Serious Adverse Events (SAEs) | Approximately up to 36 weeks
  Number of participants with SAEs will be reported. An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important, and may jeopardize participant or may require medical or surgical intervention to prevent one of the outcomes listed above.
Number of Participants Discontinued due to AEs | Approximately up to 36 weeks
  Number of participants discontinued from vaccinations or from the study due to AEs will be reported.

SECONDARY OUTCOMES:
Percentage of Participants with Seroprotection | 28 days after the third vaccination
  Percentage of participants with seroprotection will be reported. Seroprotection is defined as having a poliovirus neutralizing antibody (NAb) titer greater than or equal to (>=)8 at 28 days after the third vaccination for each poliovirus strain against Salk virus neutralization assay (VNA).
Percentage of Participants with Seroconversion | 28 days after the third vaccination
  Percentage of participants with seroconversion will be reported. Seroconversion is defined as: 1) Pre-vaccination poliovirus NAb titer less than (<)8 and post-vaccination NAb >=8 at 28 days after the third vaccination for each poliovirus strain against Salk VNA, or 2) Pre-vaccination poliovirus NAb titer >=8 and post vaccination >=4 fold increase in poliovirus NAb titer (with correction for maternal-antibody decline at Week 18, with a half-life of maternal antibodies of 1 month), at 28 days after the third vaccination for each poliovirus strain against Salk VNA.
Poliovirus Type- and Strain-specific Neutralizing Antibody (NAb) Responses | 28 days after the third vaccination
  Poliovirus NAb titers will be determined against the wild-type Salk strains (Type 1 [Mahoney], Type 2 [MEF-1] and Type 3 [Saukett]) as well as against the Sabin strains (Types 1, 2 and 3), in accordance with the World Health Organization (WHO) recommendations for immunogenicity assessment of inactivated poliovirus vaccine (IPV).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (3):
- Philippines (3):
  - De La Salle Health Sciences Institute- DLSUMC, Dasmariñas
  - De La Salle University Medical Center, Dasmariñas
  - Philippine General Hospital, Manila